CLINICAL TRIAL: NCT03376958
Title: Apatinib for Relapsed and Refractory Difuse Large B Cell Lymphoma: an Open-label, Single Armed, Exploratory Study
Brief Title: Apatinib for Relapsed and Refractory Diffuse Large B Cell Lymphoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhengzhou University (Other)
Responsible Party: Principal Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital, Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx2017-1
Record Dates: First submitted 2017-10-27; First posted 2017-12-19 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Relapsed and Refractory; Diffuse Large B Cell Lymphoma
Keywords: R R DLBCL; ORR; PFS; OS
MeSH Terms: conditions — Recurrence; Lymphoma, Large B-Cell, Diffuse | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib (Experimental): Apatinib 500mg once daily makes an initial dose and 28 days made one treatment cycle. All patients took the drug continuously until disease progression, intolerable toxicities, and patient-requested withdrawal. Appropriate supportive care were given.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib, a novel small molecule vascular endothelial growth factor receptor-2 (VEGFR-2) tyrosine kinase inhibitor, have shown remarkable efficacy in many solid cancers. The result of our study presented that apatinib might have a rapid, safe and high efficacy on lymphoma patients.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Apatinib for patients with Relapsed Refractory Diffuse Large B Cell Lymphoma.

DETAILED DESCRIPTION:
Patients with relapsed /refractory diffuse large B cell lymphoma usually have a bad prognosis. These patients cannot be treated successfully with the conventional chemotherapy of CHOP. Apatinib is a new type of oral tyrosine kinase inhibitor targeting VEGFR-2.The investigators have been proceeding this trial to evaluate the efficacy and safety of Apatinib in the patients with relapsed refractory diffuse large B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Age range 14-70 years old; ECOG performance status 0-2.
* Estimated survival time > 6 months.
* Histological confirmed diffuse large B cell lymphoma.
* Have taken first-line chemotherapy regimen and failed.
* None of chemotherapy contraindication: hemoglobin ≥ 90 g/dl, neutrophil ≥ 1.5×109/L, platelet ≥ 100×109/L, ALT and AST ≤ 2×ULN, serum bilirubin ≤ 1.5×ULN, serum creatine ≤ 1.5×upper limitation of normal (ULN), Serum Albumin ≥ 30g/L, serum plasminogen is normal.
* At least one measurable lesion.
* None of other serious diseases, cardiopulmonary function is normal.
* Pregnancy test of women at reproductive age must be negative.
* Patients could be followed up.
* None of other relative treatments including the traditional Chinese medicine, immunotherapy, biotherapy except anti-bone metastasis therapy and other symptomatic treatments.
* Volunteers who signed informed consent.

Exclusion Criteria:

* Disagreement on blood sample collection.
* Patients allergic of any of drug in this regimen or with metabolic disorder.
* Pregnant or lactating women.
* Serious medical illness likely to interfere with participation.
* Serious infection.
* Primitive or secondary tumors of central nervous system.
* Chemotherapy or radiotherapy contraindication.
* The evidence of CNS metastasis.
* History of peripheral nervous disorder or dysphrenia.
* Patients participating in other clinical trials.
* Patients taking other antitumor drugs.
* Patients estimated to be unsuitable by investigator.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | up to end of follow-up-phase
  The proportion of patients whose tumor volume has reduced to a predetermined value and can maintain the minimum time limit is the sum of complete and partial mitigation.

SECONDARY OUTCOMES:
Progression-free Survival | up to end of follow-up-phase
  The time between the start of randomization and the progression of the tumor (any aspect) or (for any reason) death
Overall Survival | up to the date of death or end of follow-up-phase
  Time from randomization to death for any reason

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Department of The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Ma X, Li L, Zhang L, Fu X, Li X, Wang X, Wu J, Sun Z, Zhang X, Feng X, Chang Y, Zhou Z, Nan F, Zhang J, Li Z, Zhang M. Apatinib in Patients with Relapsed or Refractory Diffuse Large B Cell Lymphoma: A Phase II, Open-Label, Single-Arm, Prospective Study. Drug Des Devel Ther. 2020 Jan 22;14:275-284. doi: 10.2147/DDDT.S227477. eCollection 2020. PMID 32158186